CLINICAL TRIAL: NCT01224431
Title: Needle-Free Jet Injection of Lidocaine for Local Anesthesia During Lumbar Puncture: A Randomized Controlled Trial
Brief Title: Needle-Free Jet Injection of Lidocaine During Lumbar Puncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phoenix Children's Hospital (Other)
Responsible Party: Principal Investigator, Blake Bulloch, MD, Phoenix Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-014
Record Dates: First submitted 2010-09-30; First posted 2010-10-20 (Estimated); Results first posted 2011-06-14 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-09

CONDITIONS: Pain
Keywords: pain; lidocaine; lumbar puncture; j-tip
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buffered lidocaine J-tip (Experimental): Needleless injection of buffered lidocaine prior to lumbar puncture versus placebo (Normal saline)
  Interventions: Drug: Buffered Lidocaine J-tip
- Normal saline J-tip (Placebo Comparator): Needleless injection of normal saline (placebo) prior to lumbar puncture versus use of buffered lidocaine
  Interventions: Drug: Buffered Lidocaine J-tip

INTERVENTIONS:
Drug: Buffered Lidocaine J-tip — All patients were administered the J-tip and randomized to either treatment with 1% lidocaine or an equivalent amount of sterile normal saline prior to lumbar puncture. Vital signs were recorded during the procedure. Facial expressions were video recorded
  Other Names: Normal Saline J-tip

SUMMARY:
Background: The J-Tip Device allows an intradermal needle-free jet injection of 1% buffered lidocaine. This study compares needle-free jet injection of lidocaine to saline in reducing pain prior to lumbar puncture in infants.

Methods: Randomized, double-blinded, placebo controlled trial involving infants, less than 3 months of age, presenting to the emergency department meeting clinical criteria for a lumbar puncture. All patients were administered the J-tip and randomized to either treatment with 1% lidocaine or an equivalent amount of sterile normal saline prior to lumbar puncture.

DETAILED DESCRIPTION:
Background: Lumbar puncture is an essential procedure in the emergency department for the evaluation of meningitis. Subcutaneous injection of lidocaine prior to lumbar puncture for local anesthesia is not a pain free procedure. The J-Tip Device allows an intradermal needle-free jet injection of 1% buffered lidocaine. This study compares needle-free jet injection of lidocaine to saline in reducing pain prior to lumbar puncture in infants.

Methods: Randomized, double-blinded, placebo controlled trial involving infants, less than 3 months of age, presenting to the emergency department meeting clinical criteria for a lumbar puncture. All patients were administered the J-tip and randomized to either treatment with 1% lidocaine or an equivalent amount of sterile normal saline prior to lumbar puncture. Vital signs were recorded during the procedure. Facial expressions as well as crying times were video recorded from start to finish. Independent reviewers assigned pain scores based on the validated Neonatal Facial Coding System with possible scores ranging from 0-5.

ELIGIBILITY:
Inclusion Criteria:

* fever in infants less than 3 months

Exclusion Criteria:

* toxic appearance, altered level of consciousness, age greater than 3 months or less than 4kg of weight

Max Age: 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Blake Bulloch, MD, Study Director — Phoenix Childrens Hospital
Locations (1):
- Blake Bulloch/PhoenixChildren's Hospital, Phoenix, Arizona, United States

REFERENCES:
- [Background] Ferayorni A, Yniguez R, Bryson M, Bulloch B. Needle-free jet injection of lidocaine for local anesthesia during lumbar puncture: a randomized controlled trial. Pediatr Emerg Care. 2012 Jul;28(7):687-90. doi: 10.1097/PEC.0b013e31825d210b. PMID 22743744

RESULTS

PARTICIPANT FLOW:
Groups:
- Needleless Injection of Buffered Lidocaine: needleless injection of buffered lidocaine prior to lumbar puncture
- Normal Saline Via Needleless Injection: needleless injection of normal saline prior to lumbar puncture
Period: Overall Study
Arm/Group | Needleless Injection of Buffered Lidocaine | Normal Saline Via Needleless Injection
Started | 30 | 30
Completed | 30 | 25
Not Completed | 0 | 5
Not completed — not randomized | 0 | 4
Not completed — no video record | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Needleless Injection of Buffered Lidocaine | Normal Saline Via Needleless Injection | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 30 | 60
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: days] — In days of age not years
  days | 48 (15) | 40 (18) | 44 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 14 | 15 | 29
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Pain, Measured as Units on a Scale
Description: Pain scores at time of needle insertion using neonatal facial coding score. The scale has five components; cry, brow bulge, eye squeeze; nasolabial fold and open month. Each component is either present or absent, with a value of 0 or 1 given. Minimum score of 0 and a maximum score of 5 possible
Time Frame: on average the first hour in emergency department at 4 time points during entire lumbar puncture procedure.
Measure: Mean (Standard Deviation); unit: units on scale, 0-5
Arm/Group | Needleless Injection of Buffered Lidocaine | Normal Saline Via Needleless Injection
Number analyzed (Participants) | 30 | 30
units on scale, 0-5 | 4.0 (1.3) | 4.8 (0.5)

2. Secondary Outcome: Length of Cry
Description: cry video recorded and measured after needle stick until pt stopped crying
Time Frame: On average the first hour in the emergency department; from needle stick to end of lumbar puncture
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Buffered Lidocaine J-tip: Buffered Lidocaine group: Pain Scores and Cry Time Between Groups
- Normal Saline J-tip: Normal Saline Group: Pain scores and cry time
Arm/Group | Buffered Lidocaine J-tip | Normal Saline J-tip
Number analyzed (Participants) | 30 | 25
seconds | 38.53 (18.63) | 48.76 (16.15)

ADVERSE EVENTS:
Groups:
- Buffered Lidacaine J-tip: Experimental: needleless injection of buffered lidocaine
- Normal Saline J-tip: Placebo Comparator: normal saline via needleless injection
Arm/Group | Buffered Lidacaine J-tip | Normal Saline J-tip
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No